CLINICAL TRIAL: NCT00005472
Title: Job Strain, Ambulatory Blood Pressure and Hypertension
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4954; R03HL055165 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2004-08

CONDITIONS: Cardiovascular Diseases; Cerebrovascular Accident; Hypertension; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Stroke; Hypertension; Heart Diseases

SUMMARY:
To analyze the association between an objective measure of "job strain" and risk of stroke, and change in ambulatory blood pressure.

DETAILED DESCRIPTION:
BACKGROUND:

Cardiovascular disease accounts for 43 percent of all deaths in the United States. Hypertension affects as many as 50 million Americans, however the causes of essential hypertension are not well known. A new CVD risk factor ("job strain") has emerged as a potential major cause of essential hypertension. By 1995, over 20 studies had found significant positive relationships between "job strain" and CVD, coronary heart disease, all-cause mortality or hypertension. "Job strain" is defined as high psychological workload demands combined with low"decision latitude". An expanded concept of "job strain" which included low workplace social support ("iso-strain") was developed and examined in the study.

Important questions remained to be answered about "job strain", CVD and hypertension. In most studies, "job strain" was only measured at one point in time, while, in fact, cumulative exposure to "job strain" was believed to be the risk factor. In addition, most studies relied on self-report measures of "job strain". Also, no studies specifically examined risk of stroke and "job strain".

DESIGN NARRATIVE:

Data from the Cornell University cohort study of Psychosocial Factors and Cardiovascular Disease and the Columbia University-Northern Manhattan Stroke Study were analyzed. The study had five specific aims, including to determine whether: blood pressure levels were associated with cumulative exposure to "job strain"; differences in blood pressure increases were associated with an objective measure of "job strain"; increased risk of stroke was associated with an objective measure of "job strain"; changes in psychological variables over time were associated with job characteristics; changes in CVD risk factors (other than hypertension) were associated with job characteristics.

Paul Landsbergis also constructed measures of cumulative exposure to "job strain" and determined their association with blood pressure, and analyzed the association between job characteristics and change in psychological variables and cardiovascular disease (CVD) risk factors.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1996-09; Study Completion 1998-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Landsbergis — Weill Medical College of Cornell University

REFERENCES:
- [Background] Friedman R, Schwartz JE, Schnall PL, Landsbergis PA, Pieper C, Gerin W, Pickering TG. Psychological variables in hypertension: relationship to casual or ambulatory blood pressure in men. Psychosom Med. 2001 Jan-Feb;63(1):19-31. doi: 10.1097/00006842-200101000-00003. PMID 11211061
- [Background] Landsbergis PA, Schnall PL, Pickering TG, Schwartz JE. Validity and reliability of a work history questionnaire derived from the Job Content Questionnaire. J Occup Environ Med. 2002 Nov;44(11):1037-47. doi: 10.1097/00043764-200211000-00010. PMID 12448355
- [Background] Landsbergis PA, Schnall PL, Pickering TG, Warren K, Schwartz JE. Lower socioeconomic status among men in relation to the association between job strain and blood pressure. Scand J Work Environ Health. 2003 Jun;29(3):206-15. doi: 10.5271/sjweh.723. PMID 12828390
- [Background] Landsbergis PA, Schnall PL, Pickering TG, Warren K, Schwartz JE. Life-course exposure to job strain and ambulatory blood pressure in men. Am J Epidemiol. 2003 Jun 1;157(11):998-1006. doi: 10.1093/aje/kwg095. PMID 12777363